CLINICAL TRIAL: NCT03070535
Title: APOE Genotype and Diet Influences on Alzheimer's Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Angela Hanson, Acting Instructor, Gerontology, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00001483
Record Dates: First submitted 2017-02-27; First posted 2017-03-03 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Alzheimer's Disease; Dementia
Keywords: APOE E4; cognition; metabolic markers; beta-amyloid
MeSH Terms: conditions — Alzheimer Disease; Dementia; Plaque, Amyloid

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receive either the LOW or HIGH meal for their first meal and will cross-over and receive the alternate meal for their next meal. Meals are on separate days.
Who Masked: Participant
Masking Description: Subject is not told which meal, HIGH or LOW, they receive at each meal visit until after they have completed the study. At the conclusion of study participation for each subject (after their second meal), they are told which of their meals was HIGH and which one was LOW.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIGH meal (Experimental): The HIGH meal is a 700 calorie breakfast style meal, with 50% total fat (25% saturated fat), 30% carbohydrates with a glycemic index of >70, and 20% protein.
  Interventions: Other: HIGH and LOW meal ingestion
- LOW meal (Experimental): The LOW meal is a 700 calorie breakfast style meal, with 25% of those calories coming from fat (5% saturated fat), 55% carbohydrate (with a glycemic index of <55), and 20% protein.
  Interventions: Other: HIGH and LOW meal ingestion

INTERVENTIONS:
Other: HIGH and LOW meal ingestion — The study will examine CSF biomarker responses to HIGH and LOW meals in 80 men and women with and without the E4 allele in a cross-over design. After an overnight fast, participants will ingest either a HIGH or LOW meal on separate days 3-5 weeks apart in random order. Three hours after meal ingestion, participants will undergo a cognitive battery, followed by spinal fluid collection. Blood samples will also be taken at 7 time points before and after meal ingestion.

SUMMARY:
This study involves the collection of cognitive and biomarker responses to HIGH and LOW meals in healthy older adults with and without the APOE E4 genotype. Subjects will eat the meal after an overnight fast, followed by cognitive testing, spinal fluid and blood collection. The HIGH meal will be a meal high in saturated fat and high glycemic index foods vs. LOW meal which will be low in saturated fat and low glycemic index foods.

DETAILED DESCRIPTION:
The purpose of this study is to examine how the risk gene for Alzheimer's disease APOE epsilon 4 (E4) influences acute cognitive responses to different types of meals. The rationale for this study is that we know that a diet high in saturated fat and high glycemic index foods (HIGH diet) is a risk factor for Alzheimer's disease (AD). However we have found paradoxically that a Western style HIGH diet acutely improved cognition in APOE E4 carriers, but worsened cognition in E4 non-carriers. This experiment will examine mechanisms that underlie this differential response between E4 carriers and non-carriers.

We will enroll older adults who do not have dementia, half of which will be E4 carriers and the other half will be non-carriers. Both groups will contain equal numbers of men and women. These individuals will undergo two experiments in which they eat either a high or a low fat meal, and then after the meal will undergo several tests. The outcome measures include blood measures of metabolic markers, cognitive tests that are known to be sensitive to changes even after a single meal, and spinal fluid measures of Alzheimer's biomarkers such as beta-amyloid, as well as spinal fluid levels of lipids, glucose and insulin. This study will allow us to test whether high and low fat meals acutely affect cognitive and Alzheimer's biomarkers, and if those changes depend on APOE genotype or gender. It is our hope that this work will contribute to our broader understanding about the risks of diet and AD, to help us understand more about how to prevent and treat this devastating neurological disease.

ELIGIBILITY:
Inclusion Criteria:

1. Written consent is signed and dated by the subject.
2. Subject is at least 55 years of age or older, and if female, must be post-menopausal for at least one year, or be one year out from a hysterectomy.
3. Able to read and understand English
4. Be free of dementia, and able to cognitively and physically give informed consent.
5. In the opinion of the investigator, the subject will be able to complete the study procedures.

   -

Exclusion Criteria:

1. Diabetes: Known type 1 or Type 2 diabetes, currently taking diabetic medications or insulin, and/or fasting blood glucose ≥ 126 as per the 2009 American Diabetes Association guidelines. Remote use of diabetic agents, or a history of gestational diabetes, is ok.
2. Liver and kidney disease: Active liver disease will be excluded. Also excluded are elevations in liver function tests of SGOT (AST) and/or SGPT (ALT) > 1.5 times the upper limit of normal. Active renal disease (Stage IV or V chronic kidney disease) will also be excluded.
3. Lipid abnormalities: Diagnosis of hyperlipidemia or hypertriglyceridemia requiring statin, bile acid resins, fibrate medications, and/or high dose niacin will be excluded, as these medications may interfere with the study outcomes. If subjects are on omega-3 fatty acids, low dose niacin, or other alternative/herbal remedies such as red yeast rice, they can be enrolled if they agree to stop the medication during the study period. Also excluded are significant cholesterol abnormalities as defined by the Adult Treatment Panel III classification: LDL cholesterol ≥190 mg/dL, total cholesterol ≥240 mg/dL, or triglycerides > 200. HDL levels outside of the typical range are ok.
4. Dementia and cognitive impairment: Known diagnosis of dementia, use of dementia medications, or identification of dementia during the baseline visit, will be excluded. Also excluded are other significant neurologic diseases which affect cognition, such as recent stroke, recent severe head injury, or advanced Parkinson's disease. Mild cognitive impairment with no functional deficits is ok.
5. Contraindications to lumbar puncture: Those with medical conditions that preclude a lumbar puncture such as an intracranial tumor, lower spinal hardware, or use of anticoagulation, will be excluded. Daily aspirin for prevention is ok. Use of NSAIDS is ok as long as participant uses them as needed rather than daily, and is able to discontinue these agents two days prior to the LP procedures.
6. Significant medical illnesses: Illnesses which would cause a hardship on the participant to attend study visits and undergo a lumbar puncture. This includes uncontrolled severe hypertension, unstable angina or cardiovascular disease, moderate pulmonary disease (COPD), and Class III-IV congestive heart failure (CHF).
7. Active malignancy undergoing treatment with chemotherapeutic or radiation treatments. Remote history of treated cancer is ok, as long as current cognition and digestion are not affected
8. Treatment with hormones: Use of estrogen, testosterone, and continuous corticosteroid replacements will be excluded, as these may have effects on study outcomes. Women must be post-menopausal for at least 1 year before enrolling in the study, or be one year out from a hysterectomy. Women who use hormone replacement therapy for symptomatic menopause can be enrolled, if they agree to discontinue the medication four weeks before the first meal and then throughout the study. Transgendered subjects can be included in the study, provided that they are not taking sex steroids.
9. Psychiatric disorders: Subjects who report active untreated major depression, psychosis, or mania, or who present with those symptoms at the baseline visit, will be excluded. Psychiatric conditions such as post-traumatic stress disorder (PTSD), depression, and anxiety which are stable and treated with medication or therapy are ok.
10. Major digestive disorders including inflammatory bowel diseases, irritable bowel syndrome, and celiac disease. History of surgical procedures which may affect the absorption of meals, such as any weight loss surgery such as gastric bypass or banding, or small intestine resection. Acid reflux is allowed if participant is on a stable medication regimen.
11. Food allergies and intolerances: Those subjects allergic to the ingredients of the meals will be excluded. Also excluded are medical conditions requiring strict adherence to a particular diet, such as celiac disease or phenylketonuria.
12. Alcohol use: While they are in the study, subjects will be asked to limit their alcohol intake to two drinks per day or less for men, or one drink per day or less for women, due to alcohol's effects on lipid biochemistry and the study outcomes. Subjects who are unable or unwilling to meet these criteria will not be enrolled.

    -

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Lipid biomarkers | 4 hours post meal
  Paired serum and cerebrospinal fluid levels of free fatty acids and triglycerides
APOE lipidation | 4 hours post meal
  Cerebrospinal fluid levels of total ApoE, and lipidated ApoE
Insulin | 4 hours post meal
  Paired serum and cerebrospinal fluid levels of insulin

CONTACTS AND LOCATIONS:
Overall Officials: Angela J Hanson, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided